CLINICAL TRIAL: NCT06367166
Title: Study of the Effects of Bioflavonoids on Venous Wall Remodeling in Patients With Varicose Veins of the Lower Extremities
Brief Title: Effects of Bioflavanoids on Vascular Wall Remodeling in Patients With Varicose Veins
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ryazan State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RyazanSMU
Record Dates: First submitted 2023-10-02; First posted 2024-04-16 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Varicose Veins of Lower Limb; Varix; Vascular Diseases; Leg Edema
Keywords: bioflavonoids; venous remodeling; varicose veins
MeSH Terms: conditions — Varicose Veins; Vascular Diseases | interventions — Diosmin; Hesperidin; Flavonoids; Fibronectins; Plasminogen Activator Inhibitor 1; Vimentin; Platelet Endothelial Cell Adhesion Molecule-1

STUDY DESIGN:
Intervention Model Description: Patients with varicose veins will be assigned to different treatments to assess the venous wall remodeling parameters throughout treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- А- Varicose vein patients with Conservative treatment with a venoactive drug (Experimental): 20 patients with varicose veins who will be treated conservatively - receive the drug "Venarus®" (diosmin in combination with hesperidin) at a dosage of 1000 mg once daily for 6 months along with elastic compression
  Interventions: Drug: "Venarus®" (diosmin and hesperidin); Other: Elastic compression; Other: Evaluation of biomarkers of venous wall remodeling (fibronectin, PAI-1, vimentin, vWF, CD31), venous symptoms and severity scores
- B- Varicose veins patients without invasive treatment or a venoactive drug (Experimental): 20 patients with varicose veins C2s-C3s who are not prescribed conservative therapy with a venoactive drug and will not undergo invasive treatment; the patients will receive elastic compression
  Interventions: Other: Elastic compression; Other: Evaluation of biomarkers of venous wall remodeling (fibronectin, PAI-1, vimentin, vWF, CD31), venous symptoms and severity scores
- C- Varicose veins patients who will undergo EVLA and conservative treatment with a venoactive drug (Experimental): 20 patients with varicose veins who will undergo invasive treatment (endovenous laser ablation with miniphlebectomy), followed by Venarus at a dosage of 1000 mg once daily for 6 months; the patients will also receive elastic compression
  Interventions: Drug: "Venarus®" (diosmin and hesperidin); Procedure: Endovenous laser ablation (EVLA) with miniphlebectomy; Other: Elastic compression; Other: Evaluation of biomarkers of venous wall remodeling (fibronectin, PAI-1, vimentin, vWF, CD31), venous symptoms and severity scores
- D- Varicose veins patients who will undergo EVLA (Experimental): 20 patients with varicose veins patients who will undergo invasive treatment (EVLK with miniphlebectomy), after which no venoactive drugs will be prescribed; the patients will also receive elastic compression
  Interventions: Procedure: Endovenous laser ablation (EVLA) with miniphlebectomy; Other: Elastic compression; Other: Evaluation of biomarkers of venous wall remodeling (fibronectin, PAI-1, vimentin, vWF, CD31), venous symptoms and severity scores
- E-healthy volunteers (Experimental): 20 healthy volunteers without clinical and ultrasound signs of varicose veins receiving no treatment
  Interventions: Other: Evaluation of biomarkers of venous wall remodeling (fibronectin, PAI-1, vimentin, vWF, CD31), venous symptoms and severity scores

INTERVENTIONS:
Drug: "Venarus®" (diosmin and hesperidin) — "Venarus®" (diosmin and hesperidin) at a dosage of 1000 mg once daily for 6 months
  Other Names: BIOFLAVANOIDS
  Arms: C- Varicose veins patients who will undergo EVLA and conservative treatment with a venoactive drug; А- Varicose vein patients with Conservative treatment with a venoactive drug
Procedure: Endovenous laser ablation (EVLA) with miniphlebectomy — Endovenous laser ablation will be performed under local and tumescent anesthesia, laser wavelength 1470nm.
  Arms: C- Varicose veins patients who will undergo EVLA and conservative treatment with a venoactive drug; D- Varicose veins patients who will undergo EVLA
Other: Elastic compression — All subject with varicose veins enrolled in the study will receive class 2 elastic compression (elastic stockings) after enrollment
  Arms: B- Varicose veins patients without invasive treatment or a venoactive drug; C- Varicose veins patients who will undergo EVLA and conservative treatment with a venoactive drug; D- Varicose veins patients who will undergo EVLA; А- Varicose vein patients with Conservative treatment with a venoactive drug
Other: Evaluation of biomarkers of venous wall remodeling (fibronectin, PAI-1, vimentin, vWF, CD31), venous symptoms and severity scores — The patients and healthy volunteers will undergo evaluation of biomarkers of venous wall remodeling (fibronectin, PAI-1, vimentin, vWF, CD31), Venous clinical severity (VCS) score, Visual Analog Scale (VAS) score and 20 item-ChronIc Venous dIsease quality-of-life Questionnaire (CIVIQ-20) at baseline, and 2, 3, and 6 months after enrollment

SUMMARY:
The study is aimed at assessing the dynamics of changes in biochemical markers of venous wall remodeling (type 1 plasminogen activation inhibitor (PAI-1), fibronectin (fibronectin, FN), vimentin (vimentin, VM), von Willebrand factor (vWF), PECAM-1 (CD31) ) in patients with C2s-C3s varicose veins compared with healthy volunteers while taking Venarus® (diosmin in combination with hesperidin).

DETAILED DESCRIPTION:
The study will include 80 patients with varicose veins of the lower extremities, CEAP (CEAP classification stands for Clinical (C), Etiological (E), Anatomical (A), and Pathophysiological (P)) clinical class C2s-C3s and 20 healthy volunteers of similar age, gender, and ethnicity (100 patients altogether). The study participants will be divided into five groups: Group A: 20 patients with varicose veins who will be treated conservatively - receive the drug "Venarus®" (diosmin in combination with hesperidin) at a dosage of 1000 mg once daily for 6 months; Group B: 20 patients with varicose veins C2s-C3s who are not prescribed conservative therapy with venoactive drugs and will not undergo invasive treatment; Group C: 20 patients with varicose veins who will undergo invasive treatment (endovenous laser ablation with miniphlebectomy), followed by Venarus at a dosage of 1000 mg once daily for 6 months; Group D: 20 patients with varicose veins who will undergo invasive treatment (endovenous laser ablation with miniphlebectomy), after which no venoactive drugs will be prescribed. Group E: 20 healthy volunteers without clinical and ultrasound signs of varicose veins.

All subjects in groups A, B, C, and D will receive elastic compression.

ELIGIBILITY:
Inclusion Criteria:

* The study will include men or women over 18 years of age with varicose disease of the lower extremities C2-C3 according to the CEAP classification, confirmed by ultrasound duplex scanning of the veins of the lower extremities

Exclusion Criteria:

* the presence of neoplasms, previous operations on the vessels of the lower extremities, deep vein thrombosis, severe concomitant diseases, including infectious ones, pregnancy, lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
changes in biomarkers of venous wall remodeling | At baseline, and at 2, 3 and 6 months after the start of treatment
  Changes in biomarkers of venous wall remodeling including vimentin, fibronectin, PAI-1, vWF, CD31
Changes in biomarkers expression in venous wall | 6 months
  Changes in expression of biomarkers of venous wall remodeling (vimentin, fibronectin, PAI-1, vWF, CD31) as assessed with Western blot techniques using the dilated veins harvested during miniphlebectomy

CONTACTS AND LOCATIONS:
Overall Officials: Igor Suchkov, Principal Investigator — RyazSMU
Locations (1):
- RyazanSMU, Ryazan, Russia